CLINICAL TRIAL: NCT04220307
Title: A Single-arm, Open-label, Multicenter, Phase II Study of AK104 in Patients With Metastatic Nasopharyngeal Carcinoma Who Have Progressed After At Least 2 Prior Lines of Chemotherapy
Brief Title: A Study of a PD-1/CTLA-4 Bispecific Antibody AK104 in Patients With Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-204
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Immuno-oncology; PD-1/CTLA-4 Bispecific
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 6 mg/kg (Experimental): AK104 IV every 2 weeks (q2w)
  Interventions: Biological: AK104
- AK104 15 mg/kg (Experimental): AK104 IV every 3 weeks (q3w)
  Interventions: Biological: AK104

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 by intravenous administration

SUMMARY:
This is a single-arm, open-label, multicenter, phase II study to evaluate the anti-tumor activity, PK and immunogenicity of AK104 in patients with metastatic nasopharyngeal carcinoma who have progressed after at least 2 prior lines of systemic chemotherapy (of which one of them must be platinum-based chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the ICF.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Expected life expectance ≥ 3 months.
* Histologically confirmed diagnosis of nonkeratinizing differentiated or undifferentiated NPC.
* Not suitable for radical local therapy.
* Stage IVb metastatic NPC patients who have failed the first-line platinum-based chemotherapy and the second-line chemotherapy.
* At least one measurable tumor lesion per RECIST 1.1 criteria. A lesion previously treated with local therapies such as radiotherapy can be considered a target lesion if there is objective evidence of progression in the lesion.
* Subjects must provide an available tumor tissue sample taken within 3 years prior to enrollment.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product

Exclusion Criteria:

* Receipt of last radiotherapy or any anti-tumor treatment [chemotherapy, targeted therapy] within 3 weeks prior to the first dose of study treatment, Receipt of last Chinese herbal drugs with antitumor indications within 1 week prior to the first dose of study treatment.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR and OX40 etc).
* Other invasive malignancies within 5 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Subjects with active autoimmune disease that requires systematic treatment in the past two years, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
* Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
* Subjects who require systemic corticosteroids (a dose equivalent to >10 mg/day prednisone) or other immunosuppressive drugs within 7days prior to the first dose of study drug.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Known history of primary immunodeficiency virus infection.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* History of gastrointestinal perforation and/ or fistula within 6 months prior to enrollment.
* Necrotic lesion(s) found by examinations within 4 weeks prior to enrollment, which, in the investigator's opinion, is at risk of massive bleeding.
* Known history of interstitial lung disease.
* Known history of active tuberculosis (TB).
* Serious infections within 4 weeks prior to the first dose of study drug, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 1000 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <1000 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Major surgery (as defined by the investigator) within 30 days prior to the first dose of study drug.
* Presence of meningeal metastasis, or active brain metastasis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria, with the exception of alopecia.
* Receipt of live attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live attenuated vaccine during the study.
* Known history of severe hypersensitivity to other monoclonal antibodies.
* Known allergic reactions to any ingredients of AK104
* Pregnant or lactating women.
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-26 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) or death from any cause (whichever occurs first)
Disease control rate (DCR) | up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
Duration of response (DoR) | up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Overall survival (OS) | up to 2 years
  OS is defined as the time from the date of first dosing to death from any cause
Incidence of treatment-emergent adverse events (TEAEs) | From the time of informed consent signed through 90 days after last dose of AK104
  An adverse event (AE) is any untoward medical occurrence or the deterioration of existing medical event in a clinical study subject administered an investigational drug, which does not necessarily have an unequivocal causal relationship with the investigational product
Observed concentrations of AK104 | From first dose of AK104 through 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No